CLINICAL TRIAL: NCT04829942
Title: Evaluation of the Effectiveness of "School Health Nursing Program" Implemented Under the Leadership of Nurse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Rasiha Güler, PhD Candidate, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: easternmediterraneanuniversity
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: School Health; Health Literacy
Keywords: school health; nursing; leadership; health literacy

STUDY DESIGN:
Intervention Model Description: "School Health Nursing Application Program", which is included in the first stage of the research, will be applied. Similarly, 30 people will be taken for the control group, and the sample size is 60 people, 30 being experimental and 30 control groups.
  In the second stage, the development of the "Child Health-Literacy Scale" will be carried out with 6458 students in the 9-11 age group who attend 4th and 5th grades of primary schools. Students will be determined by simple random sampling method among 4th and 5th grade students of primary schools in Kyrenia, Nicosia, Güzelyurt, Famagusta and İskele districts.
Masking Description: There will be 4th grade students of two primary schools in the Kyrenia region. In the study, it is expected that there will be a moderate increase in the scale scores of the experimental group children after the education.Similarly, 30 people will be taken for the control group, and the sample size is 60 people, 30 being experimental and 30 control groups.In the second stage, the development of the "Child Health-Literacy Scale" will be carried out with 6458 students in the 9-11 age group attending 4th and 5th grades of primary schools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): A 12-week training program will be applied to the experimental group. Pre-tests will be applied before the trainings begin, and height and weight measurement, nutrition, health perception and behavior scale and physical activity scale will be applied to the experimental group and the control group within the 3rd and 6th month after the training program begins. Scale applications will be applied within 2 days, taking into account the attention span of the students.
  Interventions: Behavioral: positive health behavior
- no intervention (No Intervention): Power point presentations will be given to the control group

INTERVENTIONS:
Behavioral: positive health behavior — Training on nutrition, physical activity, first aid, individual hygiene, violence and bullying will be provided to the initiative group.
  Arms: experimental

SUMMARY:
It is very important for children to take their own health responsibilities in giving them positive health behavior. The rapid advancement of technology, cultural differences, changing living conditions, and increasing chronic diseases show us that people should have the authority to make decisions about their own health, starting from primary school and childhood. All these bring the concept of health literacy to the fore. According to WHO, the concept of health literacy is the cognitive and social skills about individuals' ability to access, understand and use information and their desires in order to protect and improve well-being in health. Providing appropriate health education for age groups is very important for the development of health literacy in children. School-based health education is necessary for health promotion in the 21st century. Studies show that children's health literacy levels are low. There are very few scales that measure health literacy in children. Although there are no school health nursing practices in Northern Cyprus, there are no training programs to develop positive health behaviors. With this study we have planned, it is aimed to implement a training program within the scope of the "School Health Nursing Program" in primary schools selected as a pilot in Northern Cyprus and to form the foundations of School health nursing in our country in line with its results. In addition, measurement tools specific to age groups are needed to measure the level of health literacy, especially in school-age children. Therefore, another purpose of this study is to evaluate the effectiveness of this program on children by implementing an education program within the scope of the "School Health Nursing Program", which will be a first in our country, and to develop the "Child Health Literacy Scale" and to make it a significant contribution to science with this scale.

DETAILED DESCRIPTION:
Today's health systems are of great importance in protecting and improving the health of children. It is very important for children to take their own health responsibilities in giving them positive health behavior. The rapid advancement of technology, cultural differences, changing living conditions, and increasing chronic diseases show us that people should have the authority to make decisions about their own health, starting from primary school and childhood. All these bring the concept of health literacy to the fore. According to WHO, the concept of health literacy is the cognitive and social skills about individuals' ability to access, understand and use information and their desires in order to protect and improve well-being in health. It is very important to provide health education appropriate to age groups for the development of health literacy in children. School-based health education is necessary for health promotion in the 21st century. In this context, school health nurses gain great importance. School health nursing is of great importance for children to acquire positive health behaviors and to take their own health responsibilities . In addition to the importance of school health nursing, it is also important to know the health literacy levels of children. Studies show that children's health literacy levels are low. There are very few scales that measure health literacy in children. There is no scale developed to measure health literacy in primary school students in the literature. Among the topics given to children in health education, nutrition, physical activity, first aid, individual hygiene, protection from accidents and prevention of violence are among the most important.

In the development of positive health behaviors, healthy nutrition and regular physical activity behaviors, the education given at school age is very important. In this sense, important responsibilities fall on school health nurses. Although there are no school health nursing practices in Northern Cyprus, there are no training programs to develop positive health behaviors. With this study we have planned, it is aimed to implement a training program within the scope of the "School Health Nursing Program" in primary schools selected as a pilot in Northern Cyprus and to form the foundations of School health nursing in our country in line with its results. In addition, measurement tools specific to age groups are needed to measure the level of health literacy, especially in school-age children. Therefore, another purpose of this study is to evaluate the effectiveness of this program on children by implementing an education program within the scope of the "School Health Nursing Program", which will be a first in our country, and to develop the "Child Health Literacy Scale" and to make it a significant contribution to science with this scale.

GOAL

This study was planned to evaluate the effectiveness of the school health nursing program administered to primary school students under the leadership of a nurse and to develop the "Child Health Literacy Scale".

MATERIALS AND METHODS

1. Type of Research

   The research will be carried out in accordance with the methodological and randomized controlled experimental research design.
2. Place and time of the research

   The research will be carried out in two stages in state primary schools affiliated to the Ministry of National Education and Culture located within the borders of the Turkish Republic of Northern Cyprus, following the approval of the Ethics Committee and institutional permissions.
3. The universe and sample of the research

The Universe of the research will be formed by the children studying in state primary schools affiliated with the Ministry of National Education and Culture of the Turkish Republic of Northern Cyprus between the dates of the research. The study, which is planned in two stages, will be studied with two sample groups.

In the first stage: 4th grade students of two primary schools in the Kyrenia region will participate in the selection of the school where the "School Health Nursing Application Program", which is included in the first stage of the research, will be applied. In the study, it is expected that there will be a moderate increase in the scale scores of the experimental group children after the education and the effect size is high (d = 0.50) according to the Cohen scale. Accordingly, the sample size required for 80% power at d = 0.50 and α = 0.05 was determined as 30 persons for the experimental group to approach the normal distribution by using G * Power 3.1.9.2 software. Similarly, 30 people will be taken for the control group, and the sample size is 60 people, 30 being experimental and 30 control groups. The experimental and control group students will be determined with the MedCalc software using the block randomization technique.

In the second stage, the development of the "Child Health-Literacy Scale" will be carried out with 6458 students in the 9-11 age group who attend 4th and 5th grades of primary schools. Students will be determined by simple random sampling method among 4th and 5th grade students of primary schools in Kyrenia, Nicosia, Güzelyurt, Famagusta and İskele districts.

ELIGIBILITY:
Inclusion Criteria:

All male and female students in the 9-11 age group in the two primary schools where the study will be conducted.

Exclusion Criteria:

All male and female students except 9-11 age group

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
With the school health nursing program to be implemented within 6 months, a moderate increase in physical activity, nutrition and health perception and behavior scale scores of students is expected. | 6 month
  power analyze
Nutrition Behavior Scale | 6 mounth
  The scale was developed to determine the nutritional consumption of children. It consists of 14 items. High scores on the scale indicate that the children are healthy.
Health Perceptions and Health Behaviors Scale in Children | 6 Mounth
  This scale was developed by Walker Sechrst and Pender to evaluate children's health perceptions and health behaviors
Physical Activity Self-Efficacy Scale for Children | 6 Mounth
  This scale was developed to evaluate the physical activity and self-efficacy levels of primary school students

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
statistical analyze
Supporting Information: SAP, CSR

REFERENCES:
- [Background] Edmundson E, Parcel GS, Perry CL, Feldman HA, Smyth M, Johnson CC, Layman A, Bachman K, Perkins T, Smith K, Stone E. The effects of the child and adolescent trial for cardiovascular health intervention on psychosocial determinants of cardiovascular disease risk behavior among third-grade students. Am J Health Promot. 1996 Jan-Feb;10(3):217-25. doi: 10.4278/0890-1171-10.3.217. PMID 10163302
- [Background] Liu Y, Tang Y, Cao ZB, Zhuang J, Zhu Z, Wu XP, Wang LJ, Cai YJ, Zhang JL, Chen PJ. Results from the China 2018 Report Card on physical activity for children and youth. J Exerc Sci Fit. 2019 Jan;17(1):3-7. doi: 10.1016/j.jesf.2018.10.002. Epub 2018 Nov 26. No abstract available. PMID 30662507
- [Background] Chen P. Physical activity, physical fitness, and body mass index in the Chinese child and adolescent populations: An update from the 2016 Physical Activity and Fitness in China-The Youth Study. J Sport Health Sci. 2017 Dec;6(4):381-383. doi: 10.1016/j.jshs.2017.09.011. Epub 2017 Sep 29. No abstract available. PMID 30356661
- [Background] Knisel E, Rupprich H, Wunram A, Bremer M, Desaive C. Promotion of Elementary School Students' Health Literacy. Int J Environ Res Public Health. 2020 Dec 21;17(24):9560. doi: 10.3390/ijerph17249560. PMID 33371224
- [Result] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262